CLINICAL TRIAL: NCT00626743
Title: Clinical Trial to Investigate the Influence of SK3530 on the Blood Pressure of Patients With Hypertension Taking Amlodipine
Brief Title: Phase I Study to Investigate the Effect on the Blood Pressure After Oral Administration of SK3530 and Amlodipine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SK3530_AMD_I_2007
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — 2-(5-(4-(2-hydroxyethyl)piperazin-1-ylsulfonyl)-2-n-propoxyphenyl)-5-ethyl-7-n-propyl-3,5-dihydro-4H-pyrrolo(3,2-d)pyrimidin-4-one dihydrochloride; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- SK3530 (Experimental): Active Drug
  Interventions: Drug: SK3530 100mg, Placebo, Amlodipine
- Placebo (Placebo Comparator): Tablet which has the same appearance and taste but doesn't contain active ingredient
  Interventions: Drug: SK3530 100mg, Placebo, Amlodipine

INTERVENTIONS:
Drug: SK3530 100mg, Placebo, Amlodipine

SUMMARY:
To assess the pharmacodynamic effects of co-administrated SK3530 (PDE5 inhibitor) and Amlodipine, phase I study in Hypertensive patient was designed.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects 19-65 years of age inclusive
* Subjects with hypertension as defined 100 mmHg ≤ SBP<140 mmHg and 65 mmHg ≤ DBP < 90 mmHg after more than 5 minutes in the supine position
* Written informed consent
* Willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Subjects with acute or chronic disease within 4 weeks of study initiation.
* Subejcts with any gastrointestinal disorders known to alter drug absorption(except appendectomy, herniotomy, etc.)
* Subjects with any clinically significant allergic disease or with a known allergy to the PDE5 inhibitors
* Subjects with clinically significant abnormalities on laboratory tests
* Subjects with orthostatic hypotension defined as a fall in systolic blood pressure of at least 20 mmHg or diastolic blood pressure of at least 10 mmHg when a person assumes a standing position
* Subjects with abnormal QTc interval(≥440ms)
* Subjects with color-blindness or weakness
* Subejcts with alcohol, drug or caffeine abuse
* Diet known to alter drug absorption, distribution, metabolism or elimination processes
* Subjects who participated in other clinical studies within 2 months before an administration
* Other subjects who are ineligible for the study at the discretion of the principle investigator or sub-investigators

Ages: 19 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae Gook Shin, MD,PhD, Principal Investigator — Inje University
Locations (2):
- South Korea (2):
  - INJE University Pusan Paik Hospital, Pusan
  - Asan Medical Center, Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- SK3530: Active Drug
  SK3530 100mg, Placebo, Amlodipine
- Placebo: Tablet which has the same appearance and taste but doesn't contain active ingredient
  SK3530 100mg, Placebo, Amlodipine
Period: Treatment Period 1
Arm/Group | SK3530 | Placebo
Started | 6 | 7
Completed | 6 | 6
Not Completed | 0 | 1
Period: Wash-out Period of 6 Days
Arm/Group | SK3530 | Placebo
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | SK3530 | Placebo
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | INJE University Pusan Paik Hospital | Asan Medical Center | Total
Number analyzed (Participants) | 8 | 5 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.63 (6.93) | 54.00 (10.56) | 50.69 (8.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Maximal Change From Baseline in Standing SBP
Time Frame: within 8 hrs after SK3530 or placebo
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine + SK3530 | Amlodipine + Placebo
Number analyzed (Participants) | 12 | 12
mmHg | -7.42 (5.60) | -4.42 (5.37)

2. Secondary Outcome: Maximal Change From Baseline in Standing DBP
Time Frame: within 8 hrs after SK3530 or placebo
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine + SK3530 | Amlodipine + Placebo
Number analyzed (Participants) | 12 | 12
mmHg | -7.17 (5.72) | -3.50 (3.37)

ADVERSE EVENTS:
Time Frame: about 6 weeks
Description: Screening visit ~ Post-study visit
Arm/Group | Amlodipine + SK3530 | Amlodipine + Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amlodipine + SK3530 (N=12) | Amlodipine + Placebo (N=12)
Dizziness (Cardiac disorders) | 0 (0) | 1 (1)
Flushing(facial flushing) (Vascular disorders) | 1 (1) | 0 (0)
Vascular Headache(headache) (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release